CLINICAL TRIAL: NCT05148468
Title: Effects of Spinal Cord Stimulation on Gait in Patients With Parkinson´s Disease; a Randomized, Crossover, Double Blinded, Placebo-Controlled Study
Brief Title: Effects of Spinal Cord Stimulation on Gait in Patients With Parkinson´s Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No effect identified with two thirds of expected sample size completing study, one patient presented adverse perioperative event.
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCSPDgait
Record Dates: First submitted 2021-11-04; First posted 2021-12-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: gait; Parkinson´s disease; Spinal Cord stimulation
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Double blinded randomized placebo controlled cross over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and examiners will be blinded to stimulation status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active stimulation (Experimental): During active stimulation phase, patients will receive through the spinal cord stimulator active tonic stimulation with amplitude set to 90% of paresthesia inducing threshold, therefore allowing blinding. Patients will be evaluated after a three week wash out period with no stimulation and after three weeks of continuous active stimulation.
  Interventions: Device: Active spinal cord stimulation
- Sham stimulation (Sham Comparator): During sham stimulation phase, patients will receive through the spinal cord stimulator a zero amplitude stimulation, therefore having no electrical current passing through epidural leads but with the program status still displayed as "on" if checked with patient's personal controller. Patients will be evaluated after a three week wash out period with no stimulation and after three weeks of continuous sham stimulation.
  Interventions: Device: Sham spinal cord stimulation

INTERVENTIONS:
Device: Active spinal cord stimulation — Spinal cord stimulation is accomplished with surgically implanted epidural leads at Th3 - Th4 levels and a pulse generator implanted in subcutaneous fat. During active stimulation amplitude will be set to 90% paresthesia inducing threshold.
  Arms: Active stimulation
Device: Sham spinal cord stimulation — Spinal cord stimulation is accomplished with surgically implanted epidural leads at Th3 - Th4 levels and a pulse generator implanted in subcutaneous fat. During sham stimulation amplitude will be set to zero.
  Arms: Sham stimulation

SUMMARY:
Spinal cord stimulation (SCS) for Parkinson´s disease (PD) has been studied for a decade but consensus on efficacy is still lacking, with the previous stimulation standard paresthesia inducing threshold hampering adequate subject blinding. Considering that tonic stimulation for pain has been shown to be efficacious for most patients on subthreshold stimulation parameters we hypothesize a similar result with it´s use on PD. The investigators aim to:

1. Produce stronger evidence on SCS efficacy for PD in regards to gait, motor scores and quality of life measures by incorporating subthreshold in a randomized cross over placebo-controlled study with a large sample.
2. Identify predictors of good response to SCS therapy by performing trans spinal magnetic stimulation (TSMS) before SCS implant and correlating the response to SCS to that of the noninvasive TSMS.
3. Better provide biomarkers of SCS therapy through functional magnetic resonance imaging and electroencephalographic mapping.

DETAILED DESCRIPTION:
Gait impairment in Parkinson´s Disease (PD) is often refractory to standard medication therapy and functional surgery options currently explored resulting in grave loss of independence and quality of life. Spinal cord stimulation (SCS) has been explored for its role in PD after enthusiastic animal studies and despite mixed initial results is currently a very promising candidate for ameliorating hard to treat gait and balance disorders.

Consensus on tonic SCS efficacy is hampered mostly due to small samples and lack of randomized controlled trials so far, and the impossibility of subject blinding due to standard stimulation settings using currents over the paresthesia inducing threshold. Some small studies already attempted subthreshold blinding and all resulted in non significant results, however with no important difference when switching to suprathreshold settings, thus raising the possibility of non responder subjects or inefficient therapy and calling for additional exploration. The investigators aim to explore the feasibility of a placebo controlled trial using subthreshold stimulation with a larger sample and produce stronger evidence on SCS efficacy for PD.

Additionally, the possibility of non responder subjects will be explored by correlating the degree of response to SCS to patient demographic characteristics including age, PD severity and cognition, gait characteristics and the degree of response to trans spinal magnetic stimulation (TSMS), a non invasive magnetic stimulation of upper thoracic spinal region, aiming to identify prognostic factors for the therapy.

Finally, functional magnetic resonance imaging and electroencephalographic mapping will be performed in order to identify biomarkers of SCS therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Parkinson´s Disease with Hoehn Yahr scale between 2,5 and 4,0
* Main complaint of balance or freezing of gait
* Score of 2 or more on subitem 3.11 of the MDS UPDRS scale concerning Freezing of Gait severity.
* Capable of informed consent

Exclusion Criteria:

* Frequent lower limb, lower back or hip pain scoring 3 or more on visual analog scale
* Uncontrolled or serious comorbidities such as uncontrolled diabetes mellitus, renal disease, anticoagulation, immunosuppression or other medical conditions that present a contraindication for SCS surgery
* Psychosis, uncontrolled depression (BDI >14) or anxiety disorder (BAI >14)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change on Timed Up and Go - Test 3 Meters (TUG-Test 3M) | 6 months
  Comparison of the change in Timed Up and Go test times between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Part III | 6 months
  Comparison of change in Unified Parkinson's Disease Rating Scale score part III between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting. MDS-PDRS part II is scored from 0 to 52 with higher scores associated with worse motor related daily activities performance. MDS-UPDRS part III is scored from 0 to 132 with higher scores associated with worse motor performance in parkinson related tests.
Parkinson's Disease Questionnaire (PDQ39) | 6 months
  Comparison of change in Parkinson's Disease Questionnaire 39 (PDQ-39) between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting. PDQ39 is score from 0 to 100%, higher values are associated with worse quality of life.
New Freezing of Gait Questionnaire (NFOG-Q) | 6 months
  Comparison of change in New Freezing of Gait Questionnaire (NFOG-Q) score between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting. NFOG-Q is scored from 0 to 28, higher values are associated with more freezing of gait.
2 minute walk test | 6 months
  Comparison of change in gait speed change in 2 minute walk test between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting. Lower values correlate with better gait speed and mobility.
Mini Balance Evaluation Systems Test (Mini-BESTest) | 6 months
  Comparison of change in Mini Balance Evaluation Systems Test (Mini-BESTest) test scores between ON-stimulation and baseline and sham-stimulation and baseline in double blinded setting. Minimum value 0 and maximum value 108. Higher value is associated with better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Background] Fuentes R, Petersson P, Nicolelis MA. Restoration of locomotive function in Parkinson's disease by spinal cord stimulation: mechanistic approach. Eur J Neurosci. 2010 Oct;32(7):1100-8. doi: 10.1111/j.1460-9568.2010.07417.x. PMID 21039949
- [Background] de Andrade EM, Ghilardi MG, Cury RG, Barbosa ER, Fuentes R, Teixeira MJ, Fonoff ET. Spinal cord stimulation for Parkinson's disease: a systematic review. Neurosurg Rev. 2016 Jan;39(1):27-35; discussion 35. doi: 10.1007/s10143-015-0651-1. Epub 2015 Jul 30. PMID 26219854
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Thevathasan W, Mazzone P, Jha A, Djamshidian A, Dileone M, Di Lazzaro V, Brown P. Spinal cord stimulation failed to relieve akinesia or restore locomotion in Parkinson disease. Neurology. 2010 Apr 20;74(16):1325-7. doi: 10.1212/WNL.0b013e3181d9ed58. No abstract available. PMID 20404313
- [Background] Fenelon G, Goujon C, Gurruchaga JM, Cesaro P, Jarraya B, Palfi S, Lefaucheur JP. Spinal cord stimulation for chronic pain improved motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2012 Feb;18(2):213-4. doi: 10.1016/j.parkreldis.2011.07.015. Epub 2011 Aug 23. No abstract available. PMID 21865071
- [Background] Santana MB, Halje P, Simplicio H, Richter U, Freire MAM, Petersson P, Fuentes R, Nicolelis MAL. Spinal cord stimulation alleviates motor deficits in a primate model of Parkinson disease. Neuron. 2014 Nov 19;84(4):716-722. doi: 10.1016/j.neuron.2014.08.061. Epub 2014 Oct 30. PMID 25447740
- [Background] Pinto de Souza C, Hamani C, Oliveira Souza C, Lopez Contreras WO, Dos Santos Ghilardi MG, Cury RG, Reis Barbosa E, Jacobsen Teixeira M, Talamoni Fonoff E. Spinal cord stimulation improves gait in patients with Parkinson's disease previously treated with deep brain stimulation. Mov Disord. 2017 Feb;32(2):278-282. doi: 10.1002/mds.26850. Epub 2016 Nov 10. PMID 27862267
- [Background] Akiyama H, Nukui S, Akamatu M, Hasegawa Y, Nishikido O, Inoue S. Effectiveness of spinal cord stimulation for painful camptocormia with Pisa syndrome in Parkinson's disease: a case report. BMC Neurol. 2017 Aug 3;17(1):148. doi: 10.1186/s12883-017-0926-y. PMID 28774283
- [Background] Samotus O, Parrent A, Jog M. Spinal Cord Stimulation Therapy for Gait Dysfunction in Advanced Parkinson's Disease Patients. Mov Disord. 2018 May;33(5):783-792. doi: 10.1002/mds.27299. Epub 2018 Feb 14. PMID 29442369
- [Background] de Lima-Pardini AC, Coelho DB, Souza CP, Souza CO, Ghilardi MGDS, Garcia T, Voos M, Milosevic M, Hamani C, Teixeira LA, Fonoff ET. Effects of spinal cord stimulation on postural control in Parkinson's disease patients with freezing of gait. Elife. 2018 Aug 2;7:e37727. doi: 10.7554/eLife.37727. PMID 30070204
- [Background] Kobayashi R, Kenji S, Taketomi A, Murakami H, Ono K, Otake H. New mode of burst spinal cord stimulation improved mental status as well as motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2018 Dec;57:82-83. doi: 10.1016/j.parkreldis.2018.07.002. Epub 2018 Jul 6. PMID 30017249
- [Background] Mazzone P, Viselli F, Ferraina S, Giamundo M, Marano M, Paoloni M, Masedu F, Capozzo A, Scarnati E. High Cervical Spinal Cord Stimulation: A One Year Follow-Up Study on Motor and Non-Motor Functions in Parkinson's Disease. Brain Sci. 2019 Apr 3;9(4):78. doi: 10.3390/brainsci9040078. PMID 30987170
- [Background] Hubsch C, D'Hardemare V, Ben Maacha M, Ziegler M, Patte-Karsenti N, Thiebaut JB, Gout O, Brandel JP. Tonic spinal cord stimulation as therapeutic option in Parkinson disease with axial symptoms: Effects on walking and quality of life. Parkinsonism Relat Disord. 2019 Jun;63:235-237. doi: 10.1016/j.parkreldis.2019.02.044. Epub 2019 Mar 2. PMID 30852148
- [Background] Chakravarthy KV, Chaturvedi R, Agari T, Iwamuro H, Reddy R, Matsui A. Single arm prospective multicenter case series on the use of burst stimulation to improve pain and motor symptoms in Parkinson's disease. Bioelectron Med. 2020 Sep 28;6:18. doi: 10.1186/s42234-020-00055-3. eCollection 2020. PMID 33005705
- [Background] Lai Y, Pan Y, Wang L, Zhang C, Sun B, Li D. Spinal Cord Stimulation with Surgical Lead Improves Pain and Gait in Parkinson's Disease after a Dislocation of Percutaneous Lead: A Case Report. Stereotact Funct Neurosurg. 2020;98(2):104-109. doi: 10.1159/000505707. Epub 2020 Feb 25. PMID 32097953
- [Background] Prasad S, Aguirre-Padilla DH, Poon YY, Kalsi-Ryan S, Lozano AM, Fasano A. Spinal Cord Stimulation for Very Advanced Parkinson's Disease: A 1-Year Prospective Trial. Mov Disord. 2020 Jun;35(6):1082-1083. doi: 10.1002/mds.28065. Epub 2020 Apr 20. No abstract available. PMID 32311155
- [Background] Cury RG, Carra RB, Capato TTC, Teixeira MJ, Barbosa ER. Spinal Cord Stimulation for Parkinson's Disease: Dynamic Habituation as a Mechanism of Failure? Mov Disord. 2020 Oct;35(10):1882-1883. doi: 10.1002/mds.28271. No abstract available. PMID 33068473
- [Background] Samotus O, Parrent A, Jog M. Long-term update of the effect of spinal cord stimulation in advanced Parkinson's disease patients. Brain Stimul. 2020 Sep-Oct;13(5):1196-1197. doi: 10.1016/j.brs.2020.06.004. Epub 2020 Jun 3. No abstract available. PMID 32504828
- [Background] Reis Menezes J, Bernhart Carra R, Aline Nunes G, da Silva Simoes J, Jacobsen Teixeira M, Paiva Duarte K, Ciampi de Andrade D, Barbosa ER, Antonio Marcolin M, Cury RG. Transcutaneous magnetic spinal cord stimulation for freezing of gait in Parkinson's disease. J Clin Neurosci. 2020 Nov;81:306-309. doi: 10.1016/j.jocn.2020.10.001. Epub 2020 Oct 20. PMID 33222935